CLINICAL TRIAL: NCT02490423
Title: Improvement in Medication Adherence Through the Implementation of Personalized Nudges
Brief Title: Improvement in Medication Adherence Through the Implementation of Personalized Nudges: the ENCOURAGE Trial
Acronym: ENCOURAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Intermountain Research and Medical Foundation (Other); CareCentra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1040522
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nudges Intervention (Active Comparator): The intervention arm will employ standard cardiovascular clinical care plus the combination of the MoBe Maps Patient Activation Platform with the Intermountain Risk Score to personalize and deliver motivational nudges to each participant.
  Interventions: Other: Nudges Intervention
- Standard of Care (No Intervention): The standard of care arm will utilize Intermountain cardiovascular clinical program care processes as they are in place today for treatment of the study subjects.

INTERVENTIONS:
Other: Nudges Intervention — The intervention arm will employ standard cardiovascular clinical care plus the combination of the MoBe Maps Patient Activation Platform with the Intermountain Risk Score to personalize and deliver motivational nudges to each participant.
  Arms: Nudges Intervention

SUMMARY:
This study will determine whether a complex, data-driven protocol for assessing patient needs and providing "nudges" (reminders to be adherent with medication prescriptions) improves adherence with cardiovascular medications. This will be accomplished by performing a 12-month clinical trial of patients with an indication for statin therapy. Participants will be randomized to either an intervention or standard-of-care arm and will be followed via passive electronic means to determine if they are adherent with medication prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Indication for statin therapy (regardless of statin use history), either: 1) the presence of coronary artery disease (CAD) (either a new diagnosis or prior diagnosis), 2) low-density lipoprotein cholesterol (LDL-C) ≥190 mg/dL, 3) the presence of diabetes and LDL-C of 70-189 mg/dL in patients aged 40- 75 years, or 4) CAD-free and diabetes-free patients aged 40-75 years who have LDL-C 70-189 mg/dL and an estimated 10-year risk of CAD ≥7.5% based on the Pooled Cohort Risk Equations (http://my.americanheart.org/professional/StatementsGuidelines/Prevention Guidelines/Prevention-Guidelines_UCM_457698_SubHomePage.jsp)
* Enrollment in a SelectHealth insurance plan
* Age ≥18 years
* Planned discharge to home

Exclusion Criteria:

* Age <18 years
* Alzheimers/Dementia
* Receipt of or expected receipt of palliative care or discharge to hospice, skilled nursing facility, inpatient rehabilitation, or long-term care facility
* Any contraindication to statin agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-02-16 (Actual)

PRIMARY OUTCOMES:
Adherence with taking prescribed statin medications. | 12 (±1) months
  Adherence will be measured by examining the passively-collected data regarding the filling and refilling of the subject's prescriptions that are available electronically through SelectHealth data and calculating the proportion of time during the followup period that each subject had medication (number of days in which the medication was available after a prescription was filled divided by the total length of the follow-up period).

SECONDARY OUTCOMES:
Adherence with taking other individual cardiovascular medications. | 12 (±1) months
  Adherence with other individual cardiovascular medications (including beta-blockers, ACE inhibitors, P2Y12 inhibitors/antiplatelets, diuretics, angiotensin receptor blockers, angiotensin-receptor neprilysin inhibitors, calcium channel blockers, vasodilators, anti-arrhythmia medications, niacin, cholesterol absorption inhibitors (ezetimibe), fibrates, digoxin, and warfarin/anticoagulants). Adherence will be measured by examining the passively-collected data regarding the filling and refilling of the subject's prescriptions that are available electronically through SelectHealth data and calculating the proportion of time during the followup period that each subject had medication (number of days in which the medication was available after a prescription was filled divided by the total length of the follow-up period).
Adherence with taking all cardiovascular medications. | 12 (±1) months
  Adherence will be measured as a composite of cardiovascular medications including statins, beta-blockers, ACE inhibitors, P2Y12 inhibitors/antiplatelets, diuretics, angiotensin receptor blockers, angiotensin-receptor neprilysin inhibitors, calcium channel blockers, vasodilators, anti-arrhythmia medications, niacin, cholesterol absorption inhibitors (ezetimibe), fibrates, digoxin, and warfarin/anticoagulants. Adherence will be measured by examining the passively-collected data regarding the filling and refilling of the subject's prescriptions that are available electronically through SelectHealth data and calculating the proportion of time during the followup period that each subject had medication (number of days in which the medication was available after a prescription was filled divided by the total length of the follow-up period).
Proportion of adherent subjects per group | 12 (±1) months
  Number of patients in each group who were adherent. Adherence will be measured by examining the passively-collected data regarding the filling and refilling of the subject's prescriptions that are available electronically through SelectHealth data and calculating the proportion of time during the follow-up period that each subject had medication (number of days in which the medication was available after a prescription was filled divided by the total length of the follow-up period).
Clinical Endpoints | 12 (±1) months
  A composite of major adverse cardiovascular events and its components, including mortality, myocardial infarction, stroke, and revascularization.
Adherence with taking individual medications at interim timepoints | 3 months, 6 months, 9 months
  Adherence will be measured for individual cardiovascular medications including statins, beta-blockers, ACE inhibitors, P2Y12 inhibitors/antiplatelets, diuretics, angiotensin receptor blockers, angiotensin-receptor neprilysin inhibitors, calcium channel blockers, vasodilators, anti-arrhythmia medications, niacin, cholesterol absorption inhibitors (ezetimibe), fibrates, digoxin, and warfarin/anticoagulants. Adherence will be measured by examining the passively-collected data regarding the filling and refilling of the subject's prescriptions that are available electronically through SelectHealth data and calculating the proportion of time during the followup period that each subject had medication (number of days in which the medication was available after a prescription was filled divided by the total length of the follow-up period).
Adherence with taking the composite of all CV medications at interim timepoints | 3 months, 6 months, 9 months
  Adherence will be measured for a composite of cardiovascular medications including statins, beta-blockers, ACE inhibitors, P2Y12 inhibitors/antiplatelets, diuretics, angiotensin receptor blockers, angiotensin-receptor neprilysin inhibitors, calcium channel blockers, vasodilators, anti-arrhythmia medications, niacin, cholesterol absorption inhibitors (ezetimibe), fibrates, digoxin, and warfarin/anticoagulants. Adherence will be measured by examining the passively-collected data regarding the filling and refilling of the subject's prescriptions that are available electronically through SelectHealth data and calculating the proportion of time during the followup period that each subject had medication (number of days in which the medication was available after a prescription was filled divided by the total length of the follow-up period).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Horne, PhD, MPH, Principal Investigator — Intermountain Medical Center; Joseph B Muhlestein, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Heart Institute, Murray, Utah, United States